CLINICAL TRIAL: NCT03813784
Title: A Randomized, Open-label, Multi-center Phase III Clinical Study To Evaluate Camrelizumab (SHR-1210) Plus Capecitabine and Oxaliplatin Followed by Sequential Treatment With Camrelizumab Plus Apatinib Mesylate in Advanced or Metastatic Gastric Cancer (GC) or Gastroesophageal Junction Cancer (GEJ) Without Prior Systemic Therapy
Brief Title: A Clinical Study To Evaluate Camrelizumab (SHR-1210) Plus Capecitabine and Oxaliplatin Followed by Sequential Treatment With Camrelizumab Plus Apatinib Mesylate in Advanced or Metastatic Gastric Cancer (GC) or Gastroesophageal Junction Cancer (GEJ) Without Prior Systemic Therapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHR-1210-III-311
Record Dates: First submitted 2019-01-20; First posted 2019-01-23 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Gastric Cancer; GastroEsophageal Cancer
Keywords: PD-1; SHR-1210
MeSH Terms: conditions — Stomach Neoplasms | interventions — camrelizumab; Capecitabine; Oxaliplatin; apatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- A (Experimental): Participants receive SHR-1210 200 mg, intravenously (IV) every 3 weeks(Q3W) plus capecitabine 1000 mg/m^2 twice daily (BID) by continous oral adminstration for 14 days, followed by a recovery period of 7 days, plus oxaliplatin 130 mg/m^2, IV q3w; for 4-6 cycles followed by SHR-1210 plus apatinib 250 mg PO qd.
  Interventions: Drug: SHR-1210; Drug: Capecitabine; Drug: Oxaliplatin; Drug: Apatinib
- B (Active Comparator): Capecitabine 1000 mg/m^2 twice daily (BID) by continous oral adminstration for 14 days, followed by a recovery period of 7 days, plus Oxaliplatin 130 mg/m^2, IV q3w
  Interventions: Drug: Capecitabine; Drug: Oxaliplatin
- C (Experimental): Participants receive SHR-1210 200 mg, intravenously (IV) every 3 weeks(Q3W) plus capecitabine 1000 mg/m^2 twice daily (BID) by continous oral adminstration for 14 days, followed by a recovery period of 7 days, plus oxaliplatin 130 mg/m^2, IV q3w; for 4-6 cycles followed by SHR-1210
  Interventions: Drug: SHR-1210; Drug: Capecitabine; Drug: Oxaliplatin

INTERVENTIONS:
Drug: SHR-1210 — Subjects receive SHR-1210 intravenously, Dosage form: lyophilised powder, Strength: 200 mg /vial
  Arms: A; C
Drug: Capecitabine — 1000 mg/m^2 administered as continuous oral twice daily (BID) of each 3-week cycle.
Drug: Oxaliplatin — 130 mg/m^2 administered IV Q3W on Day 1 of each 3-week cycle.
Drug: Apatinib — 250 mg administered as continuous oral once daily (QD) of each 3-week cycle.
  Arms: A

SUMMARY:
This is a randomized, open-label, multi-center, phase III trial to evaluate the efficacy and safety of SHR-1210 plus capecitabine and oxaliplatin sequenced by SHR-1210 plus apatinib versus capecitabine and oxaliplatin as first-line therapy in patients with locally advanced or metastatic gastric or gastroesophageal junction (GEJ) adenocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Has histologically- or cytologically-confirmed diagnosis of locally advanced unresectable or mestastatic adenocarcinoma of stomach or the esophagogastric junction (GEJ)
* Age ≥ 18 years old, male or female
* NO previous therapy for advanced/metastatic disease of GC/GEJ (including HER-2 inhibitor). Subjects with previous adjuvant/neo-adjuvant therapy completed more than 6 months can be enrolled.
* Has measurable disease per RECIST 1.1
* Eastern Cooperative Group (ECOG) performance status of 0 to 1
* Has adequate organ function
* Females of childbearing potential (FOCBP), who are not surgically sterile or postmenopausal, must conduct pregnancy test (serum or urine) within 7 days before enrollment, and must not be pregnant or breast-feeding women. If the result is negative, she must agree to use adequate contraception during the experiment and 3 months after the last administration of the test drugs. And non-sterilized males who are sexually active must agree to use adequate contraception during the experiment and 3 months after the last administration of the test drugs.

Exclusion Criteria:

* Has known HER2-positive status
* Has known active central nervous system metastatases
* Has received a live vaccine within 4 weeks prior to the first dose of study treatment
* With any acitve autoimmune disease or history of autoimmune disease, including but not limited to the following: hepatititis, pneumonitis, uveitis, colitis (inflammatory bowel disease), hypophysitis, vasculitis, nephritis, hyperthyroidism, and hypothyroidism, except for subjects with vitiligo or resolved childhood asthma/atopy. Asthma that requires intermittent use of bronchodilators or other medical intervention should also be excluded.
* Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-CTLA-4 antibody, or a VEGFR inhibitor.
* Clinically significant cardiovascular and cerebrovascular diseases, including but not limited to severe acute myocardial infarction within 6 months before enrollment, unstable or severe angina, Congestive heart failure (New York heart association (NYHA) class > 2), orventricular arrhythmia which need medical intervention.
* Hypertension and unable to be controlled within normal level following treatment of anti-hypertension agents: systolic blood pressure > 140 mmHg, diastolic blood pressure > 90 mmHg.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 885 (Actual)
Dates: Start 2019-03-07 (Actual); Primary Completion 2023-06-07 (Actual); Study Completion 2023-06-07 (Actual)

PRIMARY OUTCOMES:
Overall survival (OS) of SHR-1210 in combination with capecitabine + oxaliplatin sequenced by SHR-1210+apatinib versus capecitabine + oxaliplatin in all subjects or programmed cell death ligand 1 (PD-L1) positive participants | Up to 36 months after the first participant is randomized.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) per Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 | Up to approximately 36 months.
Progression-free Survival (PFS) per RECIST 1.1 | Up to approximately 36 months.
Incidence and severity of adverse events (AEs) | Up to approximately 36 months.
Incidence and severity of serious adverse events (SAEs) | Up to approximately 36 months.
Overall survival (OS) rates at 12 months, 18 months and 24 months | Up to approximately 12 months, 18 months and 24 months.
Progression-free Survival (PFS) rates at 6 months | Up to approximately 6 months.
Disease Control Rate (DCR) per RECIST 1.1 | Up to approximately 36 months.
Duration of Response (DoR) per RECIST 1.1 | Up to approximately 36 months.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Cancer Hospital, Peking University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided